CLINICAL TRIAL: NCT00557297
Title: NIS for Patients Using Symbicort Turbuhaler for Maintenance and Reliever Therapy in a Single Inhaler
Acronym: SYMCO
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: D5890L00031
Record Dates: First submitted 2007-11-09; First posted 2007-11-14 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Asthma
Keywords: asthma; SMART; inhaled; glucocorticosteroid; reliever; maintenance; single inhaler
MeSH Terms: conditions — Asthma; Respiratory Aspiration

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this non-interventional study is to ensure that patients in routine clinical practice follow given treatment instructions and to evaluate the number of reliever inhalations as well as the number of patient/days with more than 8/12 total inhalations at any day. If the number of reliever inhalations and thus the received inhaled glucocorticosteroid dose is not excessive, the safety conclusions from the clinical studies can be extrapolated to real life for better acceptance of SMART (Symbicort Maintenance and Reliever Therapy).

ELIGIBILITY:
Inclusion Criteria:

* Persistent asthma
* Prior Symbicort Turbuhaler maintenance and reliever therapy in a single inhaler

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2007-10; Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- Latvia (22):
  - Research Site, Alūksne
  - Research Site, Aozkraukle
  - Research Site, Balvi
  - Research Site, Cēsis
  - Research Site, Gulbene
  - Research Site, Jēkabpils
  - Research Site, Jumprava
  - Research Site, Krāslava
  - Research Site, Kuldīga
  - Research Site, Ķekava
  - Research Site, Liepāja
  - Research Site, Limbaži
  - Research Site, Līvāni
  - Research Site, Madona
  - Research Site, Ogre
  - Research Site, Preiļi
  - Research Site, Rēzekne
  - Research Site, Salacgrīva
  - Research Site, Saldus
  - Research Site, Talsi
  - Research Site, Valniera
  - Research Site, Ventspils